CLINICAL TRIAL: NCT04779463
Title: Role of Ultrasound Assessment of Parasternal Intercostal Muscle Thickness During Weaning From Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wesameldin Abelrahman Soltan (Other)
Responsible Party: Sponsor-Investigator, Wesameldin Abelrahman Soltan, Associate Professor, Menoufia University
Organization: Menoufia University (Other)
Other Study IDs: Parasternal Intercostals US
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Parasternal Intercostal Muscle Thickness; Weaning From Mechanical Ventilation
Keywords: mechanical ventilation, parasternal muscle thickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical Ventilated patients: All patients are invasively mechanically ventilated at least 24 hours, and are clinically stable as ready to undergo a spontaneous breathing trial.
  Interventions: Diagnostic Test: Parasternal intercostal muscles thickness ultrasound indicies

INTERVENTIONS:
Diagnostic Test: Parasternal intercostal muscles thickness ultrasound indicies — Parasternal intercostal muscles thickness ultrasound indicies includes:
  * Parasternal Intercostals Thickness Fraction.
  * Parasternal Intercostals Thickness at the End of Inspiration.
  * Parasternal Intercostals thickness at the End of Expiration.
  Other Names: Diaphragmatic thickness

SUMMARY:
Assessment of the the parasternal intercostal muscles thickness by the ultrasonography as a weaning predictor of the mechanically ventilated patients

DETAILED DESCRIPTION:
impact of parasternal muscle thickness on the weaning process of the mechanically ventilated patients in ICU

ELIGIBILITY:
Inclusion Criteria:

Any patient invasively mechanically ventilated at least 24 hours on a pressure support mode who is clinically stable and ready to undergo a spontaneous breathing trial.

All patients will be:

* Alert.
* Afebrile.
* Adequate cough with absence of excessive tracheobronchial secretion.
* Fraction of inspired oxygen (FIO2) of <50%.
* PEEP ≤8 cmH2O.
* PaO2/FiO2 > 150.
* pH ≥7.35 and ≤7.45.
* Respiratory rate (RR) ≤35 breaths/min.
* Hemodynamically stable in the absence of vasopressors.
* Stable metabolic and endocrinal status.
* Euglycemic state.
* Adequate mentation (no sedation or stable neurologic patient).

Exclusion Criteria:

Diaphragmatic paralysis (detected by ultrasonography).Patients&Methods. 6

* Pregnant women.
* Age: >= 18 years.
* Surgical dressings over measurement point which would preclude ultrasound exam.
* Underweight patients (Body mass index <18.5 kg/m2).
* Morbidly obese patient (Body mass index ≥ 40 kg/m2).
* Primary neuro-muscular diseases.
* Central coditions with depressed central respiratory drive (encephalitis, and brainstem haemorrhage/ischaemia).
* Repiratory conditions with reduced pulmonary compliance (interstitial lung disease, pulmonary hemorrhage, and diffuse pulmonary infiltrates) or reduced chest wall compliance (kyphoscoliosis).
* Cardiac conditions with high risk of weaning induced pulmonary edema (congestive heart failure, cyanotic heart diease, pulmonary hypertension, and ischemic heart diease).
* Addict patients.
* Patients with psychiatric disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are invasively mechanically ventilated at least 24 hours, and are clinically stable as ready to undergo a spontaneous breathing trial (SBT).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
the thickness fraction of the parasternal intercostal muscle as a predictor of successful spontaneous breathing trials | Before the start spontaneous breathing trial
  The primary outcome is to assess the change of the parasternal intercostal muscles thickness at end of expiration and end of inspiration to verify the thickness fraction of the parasternal intercostal muscle as a predictor of successful spontaneous breathing trials.

CONTACTS AND LOCATIONS:
Overall Officials: Wesameldin A Soltan, M.D., Study Director — faculty of medicine, Menoufia University
Locations (1):
- Faculty of Medicine - Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided